CLINICAL TRIAL: NCT01991600
Title: A Pilot Study to Assess the Influence of Dietary Organic Acids on Iron Absorption.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, dora pereira, Dr, Medical Research Council
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 6129
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Iron Deficiency Anaemia
Keywords: iron absorption; bioavailability; anaemia; iron deficiency; ferrous sulphate
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous Sulphate (Active Comparator): The active comparator was the standard-of-care therapy for iron deficiency anaemia (namely ferrous sulphate). Generic uncoated ferrous sulphate tablets BP 300 mg containing 60mg elemental iron were purchased from a local pharmacy. The route of administration was oral. Each participant ingested one ferrous sulphate tablet (60 mg Fe) on one of the study visits.
  Interventions: Dietary Supplement: ferrous sulphate
- ferric iron oxide-organic acid (Fe-OA) (Experimental): Fifteen different ferric iron oxide-organic acid preparations were investigated. Most organic acids used were generally recognised as safe (GRAS) and all were used at dietary equivalent levels. The dosage was 58 ± 6 mg elemental iron equivalent (average of all compounds). The route of administration was oral using methyl-cellulose capsules. On one of the study visits, each participant ingested a single dose, equivalent to ca. 60 mg iron, of the Fe-OA preparation allocated to her.
  Interventions: Dietary Supplement: ferric iron oxide-organic acid (Fe-OA)

INTERVENTIONS:
Dietary Supplement: ferrous sulphate
  Arms: Ferrous Sulphate
Dietary Supplement: ferric iron oxide-organic acid (Fe-OA)
  Arms: ferric iron oxide-organic acid (Fe-OA)

SUMMARY:
Iron deficiency is the most common micronutrient deficiency in the world today, affecting more than 60% of the global population (www.who.int/nut/ida.htm). The two main strategies for the prevention and treatment of iron deficiency involve fortification of food with iron, or direct supplementation with iron tablets. Simple iron salts (e.g. ferrous sulphate) are well absorbed but at supplemental levels (and potentially at lower levels, as used in food fortificants) can induce free radical activity resulting in gastrointestinal side effects and systematic oxidative stress. As a result, supplementation has poor compliance and improvement in iron status is compromised. Ferric salts are less inclined to produce side effects and although they are relatively well absorbed at fortification levels in food, they are poorly absorbed at the higher supplemental doses. Because certain components of food, such as organic acids, can facilitate ferric iron absorption, we now wish to determine whether dietary organic acids may similarly enable efficient absorption of supplemental ferric iron while preventing the formation of non-transferrin-bound iron (NTBI) which is a proxy for free radical activity. Our strategy is to use an iterative process between in vitro and in vivo experimentation, aimed at identifying the best choice of organic acid and the optimal ratio of iron:organic acid. The study was a cross-over, single-dose comparison against standard-of-care therapy (namely ferrous sulphate) in mildly iron deficient anaemic women. Both the investigational products and the active comparator were administered as a single dose on 2 different occasions, i.e. the investigational products on the first study visit and the active comparator 14 days later on the second study visit.

DETAILED DESCRIPTION:
The study was a first-in-human iron absorption study of ferric iron oxide-organic acid preparations (Fe-OAs). The study design was cross-over, single-dose, single-blinded comparison against standard-of-care therapy (namely ferrous sulphate) in mildly iron deficient anaemic women. Methyl-cellulose capsules containing single doses of Fe-OAs (60 mg elemental iron equivalent) were given to four subjects per test mixture to determine iron absorption and bioavailability. The study was initially designed in 2 parts (A and B). Part A was an iterative process to determine the best choice of organic acids and the optimal ratio of iron to organic acid that allowed efficient iron absorption, while part B was a comparison of absorption of the two most promising Fe-OA preparations against the standard-of-care therapy (namely ferrous sulphate). Following this iterative-based study we had a candidate Fe-OA preparation that showed nearly equivalent bioavailability to ferrous sulphate and we decided to stop the study at the end of Part A.

On day 1 of the study (Part A), the participants were given one methyl-cellulose capsule containing one of the Fe-OA preparations to be taken on an empty stomach or with a light breakfast consisting of water and 2 slices of white bread with jam. Participants were blinded to which test preparation they received. Serial serum iron levels were obtained at baseline and then 30, 60, 90, 120, 180, 210 and 240 minutes after ingestion of the iron dosage. Fourteen days later the participants returned for the second study visit where they ingested one ferrous sulphate tablet with a light breakfast, and the same visit protocol was followed. Each subject acted as her own control.

The bioavailability of iron from the Fe-OA preparations was determined by measuring erythrocyte incorporation of labelled iron 14 days following a single oral dose. Each Fe-OA preparation was labelled with 2 mg of the stable isotope 58Fe per single dose of the Fe-OA material. Ferrous sulphate was used as a reference for oral iron therapy and to determine individuals who were non-iron absorbers. Non-iron absorbers were defined as those who had no significant net area under the curve (AUC) for serum iron following ferrous sulphate oral ingestion (i.e. this was defined as a serum iron increase ≤ 5 μM). The data obtained for these individuals were excluded from the final analysis.

The bioavailability of ferrous sulphate was determined using short-term changes in serum iron levels using published algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-45 years.

Low iron stores based on one of the following criteria:

(I) Mild iron deficiency anaemia defined as haemoglobin between 10-11.9 g/dL plus either a serum ferritin less than 20 μg/L or transferrin saturation < 10% or (II) iron deficiency defined as a serum ferritin less than 12 μg/L.

Exclusion Criteria:

* pregnancy and lactation
* surgery in the past three months
* cancer in last ten years
* known chronic infection
* chronic inflammation
* moderate or severe anaemia
* known cardiovascular disease
* chronic respiratory disease.
* history of hereditary haemochromatosis or haemoglobinopathies
* current proton pump inhibitor medication
* blood donation/heavy blood loss in the last 3 months
* iron supplementation in the past 1 month
* chronic liver disease
* renal disease
* Coeliac Disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Iron Bioavailability | 14 days
  The primary outcome was bioavailability of iron from ferric iron oxide-organic acid preparations (Fe-OA) as measured by erythrocyte incorporation of labelled iron (58Fe).

SECONDARY OUTCOMES:
Iron absorption | 4 hours
  The secondary outcomes were total iron absorption and the rates of iron absorption in the 4 hours following the ingestion of the ferric iron oxide-organic acid preparations (Fe-OA)and the active comparator (namely ferrous sulphate).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Powell, PhD, Study Chair — Medical Research Council
Locations (1):
- MRC Human Nutrition Research, Cambridge, Cambridgeshire, United Kingdom